CLINICAL TRIAL: NCT01716169
Title: Treatment of Chronic and Non-Chronic Wounds in Patients With Recessive Dystrophic Epidermolysis Bullosa Using Helicoll Collagen Dressings Versus Standard of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alfred Lane, Professor of Dermatology and Pediatrics, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24915
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Helicoll (Experimental): Helicoll will be applied to one chronic wound (approximately 6 months or more duration).
  Wound designations of "control" or "Helicoll" were placed in a sealed envelope prior to study start. When a subject was enrolled, wounds were identified as "A" or "B". Then the envelope was opened which designated whether A or B would receive control or Helicoll.
  Interventions: Device: Helicoll; Device: Standard of Care Dressings

INTERVENTIONS:
Device: Helicoll — Helicoll Collagen I Wound Dressing
Device: Standard of Care Dressings — Standard of Care wound dressings (e.g. Vaseline gauze)

SUMMARY:
The purpose of this study is to test the effectiveness of Helicoll (a collagen wound dressing) in treating chronic and non-chronic wounds of recessive dystrophic epidermolysis bullosa (RDEB) patients. Helicoll will be compared to standard wound dressings.

ELIGIBILITY:
Inclusion criteria:

1. Written consent must be obtained from subjects over age 18, or from a parent or legally authorized representative if subject is under 18. Assent will be obtained from subjects age 7 - 17.
2. Subjects with a clinical diagnosis of RDEB by a dermatologist.
3. Have at least three target wounds that meet the following criteria:

   * One chronic wound, of approximately 6 months or more duration. If the subject has an additional chronic wound of similar size and duration, this additional wound will be treated with standard dressings and followed in the study. A wound in an area that consistently heals and then breaks down again will be considered a chronic wound.
   * Two non-chronic wounds, of approximately 3 months or less duration, of similar size, and able to be dressed separately. Both wounds should have approximately the same duration.

   All wounds must be:
   * Open, and not scabbed or crusted over
   * Not actively infected
   * Not requiring surgical intervention
4. A parent or legally authorized representative must be willing and able to ensure subject is present for all required study visits (for minor subjects).
5. The subject or caregiver (or a parent or legally authorized representative for subjects under 18) must be able to follow instructions.
6. Subject must be age 7 or older.

Exclusion criteria:

1. Inability to travel to Stanford for study visits.
2. Complicating illness as determined by study investigators to be exclusionary including any infection requiring systemic antibiotics.
3. Presence or history of squamous cell carcinoma at target wound site.
4. Known bovine (cow) or ovine (sheep) sensitivity.
5. Therapy with an investigational agent during the study.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Lane, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from EB Clinic patients, organization website
Groups:
- Helicoll - Chronic Wound: Helicoll will be applied to one chronic wound (approximately 6 months or more duration)
  Helicoll: Helicoll Collagen I Wound Dressing
Period: Overall Study
Arm/Group | Helicoll - Chronic Wound
Started | 10
Standard of Care Dressings Used | 7
Completed | 6
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — inconsistent dressing application | 1

BASELINE CHARACTERISTICS:
Arm/Group | Helicoll - Chronic Wound
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.6 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Wound Surface Area Change From Baseline to Week 8
Description: Change was assessed in terms of wound surface area, as measured using the ARANZ camera. Week 8 surface area measurement was compared to baseline surface area measurement and percentage in size change was calculated.
Time Frame: Baseline and Week 8
Measure: Mean (95% Confidence Interval); unit: percentage of wound surface area
Groups:
- Standard of Care Dressing - Chronic Wound: Standard of Care dressings will be applied to one chronic wound
Arm/Group | Helicoll - Chronic Wound | Standard of Care Dressing - Chronic Wound
Number analyzed (Participants) | 3 | 3
percentage of wound surface area | -63 [-99.1 to -26.9] | -8.1 [-34.4 to 18.1]

ADVERSE EVENTS:
Groups:
- Standard of Care - Chronic Wound: Standard of Care wound dressings (e.g. Vaseline gauze) will be applied to one chronic wound (of approximately 6 months duration) if the subject has more than one chronic wound of approximately the same size and duration as Helicoll chronic wound.
Arm/Group | Helicoll - Chronic Wound | Standard of Care - Chronic Wound
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 1/10 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Helicoll - Chronic Wound (N=10) | Standard of Care - Chronic Wound (N=7)
wound infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No